CLINICAL TRIAL: NCT04216914
Title: Bone Age Study In Children (BASIC): A Simple Intervention to Improve the Quality of Bone Age X-rays
Brief Title: BASIC Study: Bone Age Study In Children
Acronym: BASIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH/13/048
Record Dates: First submitted 2015-04-23; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Skeletal Age Maturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of hand outline for bone age xray (Experimental): Where children and young people are having left hand X-rays for clinical purposes the radiographer will place a template under their hand. The plate is designed not to show up on the X-ray and to not interfere with the X-ray itself. They will be asked to match their hand to the hand outline on the template.
  Interventions: Device: Hand outline

INTERVENTIONS:
Device: Hand outline — A simple outline of a hand, to which the child tried to match their own hand on order to improve positioning.

SUMMARY:
This study will see if the introduction of a hand outline on the Xray plate on which the child rests their hand will improve the quality of the Xray and reduce exposure to additional radiation by not having xrays repeated. The child will be asked to stretch their hand flat to match the outline, thus ensuring the correct position.

DETAILED DESCRIPTION:
The study of left wrist/hand Xrays can help children's doctors to ascertain the age of a child's skeleton, know how much growing they still have to do and predict how tall they will be as an adult. The Xray requires the child to keep their hand flat and still and in the correct orientation. Some children, especially young ones, find this difficult and therefore the quality of the Xray can mean that aging the skeleton is difficult and may require the Xray to be taken again.

This study will see if the introduction of a hand outline on the Xray plate on which the child rests their hand will improve the quality of the Xray and reduce exposure to additional radiation by not having xrays repeated. The child will be asked to stretch their hand flat to match the outline, thus ensuring the correct position.

ELIGIBILITY:
Inclusion Criteria:

* Children who are having a bone age Xray as part of their endocrinological hospital management.

Exclusion Criteria:

* Patients who do not give informed consent to be included in the study.
* As this study is very small and non externally funded, we will not be able to produce translations of the information sheets and consent/assent forms. This means that where patients are unable to fully give informed consent due to language barriers, they will be excluded from the study.
* )Any child with a left hand abnormality making them unable to place their hand flat e.g. contractures will be excluded.
* Any child too young or with significant enough learning difficulties making their compliance with the instructions too problematic. This will be at the discretion of the medical professional consenting the patient and the radiographer.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in X-ray quality score with use of hand outline for TW3 x-rays | 16 months
  Will providing a radiolucent hand outline, to help children correctly position their hand whilst having a bone aging X-ray taken.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Elder, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

IPD SHARING:
Plan to Share IPD: No